CLINICAL TRIAL: NCT02110420
Title: A Phase 1, Randomized, Two-part Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of CC-90001 in Healthy Subjects
Brief Title: First-in-human Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of CC-90001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Celgene (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: CC-90001-CP-001
Record Dates: First submitted 2014-02-12; First posted 2014-04-10 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Volunteers
Keywords: Safety; Pharmacokinetics; Healthy Subjects; First-in-Human
MeSH Terms: interventions — CC-90001

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (14):
- CC-90001 10mg (Single Dose) (Experimental)
  Interventions: Drug: CC-90001
- CC-90001 30mg (Single Dose) (Experimental)
  Interventions: Drug: CC-90001
- CC-90001 60mg (Single Dose) (Experimental)
  Interventions: Drug: CC-90001
- CC-90001 120mg (Single Dose) (Experimental)
  Interventions: Drug: CC-90001
- CC-90001 240mg (Single Dose) (Experimental)
  Interventions: Drug: CC-90001
- CC-90001 10mg (Multiple Doses) (Experimental)
  Interventions: Drug: CC-90001
- CC-90001 30mg (Multiple Doses) (Experimental)
  Interventions: Drug: CC-90001
- CC-90001 60mg (Multiple Doses) (Experimental)
  Interventions: Drug: CC-90001
- CC-90001 120mg (Multiple Doses) (Experimental)
  Interventions: Drug: CC-90001
- CC-90001 240mg (Multiple Doses) (Experimental)
  Interventions: Drug: CC-90001
- Placebo (Experimental)
  Interventions: Drug: Placebo
- CC-90001 480mg (single dose) (Experimental): CC-90001 480mg will be administered as a single oral dose
  Interventions: Drug: CC-90001
- CC-90001 720mg (single dose) (Experimental): CC-90001 720mg will be administered as a single oral dose
  Interventions: Drug: CC-90001
- CC-90001 480mg (multiple doses) (Experimental): CC-90001 480mg will be administered daily for 14 days
  Interventions: Drug: CC-90001

INTERVENTIONS:
Drug: CC-90001 — CC-90001 10mg will be administered as a single dose
  Arms: CC-90001 10mg (Single Dose)
Drug: CC-90001 — CC-90001 30mg will be administered as a single dose
  Arms: CC-90001 30mg (Single Dose)
Drug: CC-90001 — CC-90001 60mg will be administered as a single dose
  Arms: CC-90001 60mg (Single Dose)
Drug: CC-90001 — CC-90001 120mg will be administered as a single dose
  Arms: CC-90001 120mg (Single Dose)
Drug: CC-90001 — CC-90001 240mg will be administered as a single dose
  Arms: CC-90001 240mg (Single Dose)
Drug: CC-90001 — CC-90001 10mg will be administered daily for 14 days
  Arms: CC-90001 10mg (Multiple Doses)
Drug: CC-90001 — CC-90001 30mg will be administered daily for 14 days
  Arms: CC-90001 30mg (Multiple Doses)
Drug: CC-90001 — CC-90001 60mg will be administered daily for 14 days
  Arms: CC-90001 60mg (Multiple Doses)
Drug: CC-90001 — CC-90001 120mg will be administered daily for 14 days
  Arms: CC-90001 120mg (Multiple Doses)
Drug: CC-90001 — CC-90001 240mg will be administered daily for 14 days
  Arms: CC-90001 240mg (Multiple Doses)
Drug: Placebo — Placebo will be administered once daily for up to 14 days depending on the Part of the study
  Arms: Placebo
Drug: CC-90001 — CC-90001 480mg will be administered as a single oral dose
  Arms: CC-90001 480mg (single dose)
Drug: CC-90001 — CC-90001 720mg will be administered as a single oral dose
  Arms: CC-90001 720mg (single dose)
Drug: CC-90001 — CC-90001 480mg will be administered daily for 14 days
  Arms: CC-90001 480mg (multiple doses)

SUMMARY:
First-in-human study to evaluate safety, tolerability, and pharmacokinetics of single and multiple ascending doses of CC-90001

DETAILED DESCRIPTION:
This is a 2-part study to be conducted at a single study center. Part 1 is a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, and pharmacokinetics of CC-90001 following a single oral dose in healthy subjects. During the course of Part 1, each subject will participate in a screening phase, a baseline phase, a treatment phase and a follow up visit. There will be a total of 7 planned cohorts, each of which will consist of a different dose level, with 8 subjects per cohort. In each cohort, 6 subjects will receive a dose of CC 90001 and 2 subjects will receive placebo depending on the randomization schedule. Administration of study drug at the next higher dose level will not begin until the safety and tolerability of the preceding dose have been evaluated and deemed acceptable by the investigator and sponsor's medical monitor. Part 2 is a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, and pharmacokinetics of CC-90001 following multiple oral doses in healthy subjects. Only doses that are safe and well tolerated in Part 1 will be administered in Part 2. During the course of Part 2, each subject will participate in a screening phase, a baseline phase, a treatment phase and a follow up visit. There will be a total of up to 6 planned cohorts, each of which will consist of a different dose level, with 8 subjects per cohort. In each cohort, 6 subjects will receive a dose of CC 90001 and 2 subjects will receive placebo depending on the randomization schedule. It is planned for study drug to be administered once daily for up to 14 days. Proposed dose levels in Part 2 may be modified and/or eliminated based on data obtained from Part 1; however, the maximum dose administered in Part 2 will not exceed the maximum tolerated dose in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* 1. Must understand and voluntarily sign a written informed consent prior to any study-related procedures being performed.

  2. Must be able to communicate with the investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules.

  3. Healthy male or female of any race between 18 to 50 years of age (inclusive) at the time of signing the informed consent, and in good health as determined by a physical examination at screening.

  4. For males: Agree to use barrier contraception not made of natural (animal) membrane [for example, latex or polyurethane condoms are acceptable]) when engaging in sexual activity with a female of childbearing potential while on study medication, and for at least 28 days after the last dose of study medication.

For females: Female subjects must have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before screening, or be postmenopausal (defined as 24 months without menses before screening, with an estradiol level of < 30 pg/mL and follicle-stimulating hormone level of > 40 IU/L at screening).

5. Must have a body mass index between 18 and 33 kg/m2 (inclusive). 6. Platelet count, absolute neutrophil count and absolute lymphocyte count must be above the lower limit of normal at the screening visit.

7. Liver function tests must be below the upper limit of normal at screening. 8. All other clinical laboratory tests must be within normal limits or acceptable to the investigator.

9. Subject must be afebrile, with supine systolic blood pressure: 90 to 140 mmHg, supine diastolic blood pressure: 50 to 90 mmHg, and pulse rate: 40 to 110 bpm at screening.

10. Must have a normal or clinically-acceptable 12-lead electrocardiogram at screening. Male subjects must have a QTcF value ≤ 430 msec. Female subjects must have a QTcF value ≤ 450 msec.

Exclusion Criteria:

* 1. History of any clinically significant and relevant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders.

  2. Any condition which places the subject at unacceptable risk if he or she were to participate in the study, or confounds the ability to interpret data from the study.

  3. Exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).

  4. Used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 30 days of the first dose administration.

  5. Used any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days of the first dose administration.

  6. Used cytochrome P450 (CYP)3A inducers and inhibitors (including St. John's Wort) within 30 days of the first dose administration.

  7. Has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism and excretion, for example, bariatric procedure. Appendectomy and cholecystectomy are acceptable.

  8. Donated blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.

  9. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual) within 2 years before dosing, or positive drug screening test reflecting consumption of illicit drugs.

  10. History of alcohol abuse (as defined by the current version of the Diagnostic and Statistical Manual) within 2 years before dosing, or positive alcohol screen.

  11. Known to have serum hepatitis or known to be a carrier of hepatitis B surface antigen or hepatitis c antibody, or have a positive result to the test for human immunodeficiency virus antibodies at screening.

  12. Smoke more than 10 cigarettes per day, or the equivalent in other tobacco products (self reported).

  13. History of ulcerative colitis, Crohn's disease, diverticular disease, any polyp(s) along the gastrointestinal tract, or colorectal cancer.

  14. History of hemorrhoids, anal fissures, rectal ulcers, minor rectal bleeding (such as red blood on toilet paper after wiping) within 5 years before the first dose administration.

  15. History of gastrointestinal bleeding or blood in stool within 5 years before the first dose administration.

  16. Any positive fecal occult blood test at screening and/or at any time prior to first dosing.

  17. Any history of constipation within 2 years before the first dose administration.

  18. Subject does not routinely have a bowel movement, at minimum, every third day.

  19. Any subject with a history of Irritable Bowel Syndrome or a history of frequent abdominal cramping, frequent diarrhea, or frequent loose stools (with frequent defined as once per week or greater).

  20. Any female subject with menses (natural or artificial). 21. Any subject taking hormonal contraception. 22. Subjects who are part of the clinical staff personnel or family members of the clinical site staff.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to 8 months overall
  Number of participants with adverse events

SECONDARY OUTCOMES:
Concentrations of CC-90001 in plasma | Up to 14 days per cohort
  Blood samples will be collected at pre-specified times to determine levels of CC-90001 in plasma
Cmax: Maximum observed plasma concentration | Up to 14 days per cohort
  Cmax will be estimated for CC-90001 using a non-compartmental approach
Tmax: Time to Cmax | Up to 14 days per cohort
  Tmax will be estimated for CC-90001 using a non-compartmental approach
AUCinf: Area under the plasma concentration-time curve from time zero extrapolated to infinity | Up to 14 days per cohort
  AUCinf will be estimated for CC-90001 using a non-compartmental approach
AUCt: Area under the plasma concentration-time curve from time zero to the last quantifiable concentration | Up to 14 days per cohort
  AUCt will be estimated for CC-90001 using a non-compartmental approach
AUCtau: Area under the plasma concentration-time curve from time zero to tau, where tau is the dosing interval | Up to 14 days per cohort
  AUCtau will be estimated for CC-90001 using a non-compartmental approach
AUCtau will be estimated for CC-90001 using a non-compartmental approach | Up to 14 days per cohort
  t1/2,z will be estimated for CC-90001 using a non-compartmental approach
CL/F: Apparent total plasma clearance when dosed orally | Up to 14 days per cohort
  CL/F will be estimated for CC-90001 using a non-compartmental approach
Vz/F: Apparent total volume of distribution when dosed orally, based on the terminal phase | Up to 14 days per cohort
  Vz/F will be estimated for CC-90001 using a non-compartmental approach
Ratio of Accumulation based on Day 1 and Day 14 AUCtau | Up to 14 days per cohort
  Ratio of accumulation will be estimated for CC-90001 using a non-compartmental approach

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weiss, MD, Study Director — Celgene Corporation
Locations (1):
- PPD Development, LP, Austin, Texas, United States